CLINICAL TRIAL: NCT00577382
Title: A Phase II Study of SU011248 in Patients With Metastatic Mucosal or Acral/Lentiginous Melanoma
Brief Title: SU011248 in Patients With Metastatic Mucosal or Acral/Lentiginous Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, F. Stephen Hodi, MD, Melanoma Disease Center Director, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-145
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Results first posted 2016-12-08 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-06

CONDITIONS: Mucosal Lentiginous Melanoma; Acral Lentiginous Malignant Melanoma
Keywords: Sutent; malignant melanoma
MeSH Terms: conditions — Melanoma | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sunitinib (Experimental): Cohort A participants received 50 mg sunitinib orally daily for 4 weeks followed by a two-week break from treatment. These 6-week cycles would be repeated until progression or unacceptable toxicity up to 1 year.
  Cohort B participants received 37.5 mg sunitinib daily on a continuous basis until progression or unacceptable toxicity up to 1 year.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib
  Other Names: Sutent; SU011248

SUMMARY:
The purpose of this study is to evaluate how effective Sunitinib works in treating acral lentiginous and mucosal melanoma which has spread beyond the local region. Suninitib is a protein-tyrosine kinase inhibitor and acts as a c-kit inhibitor drug. It is believed to work by blocking signals on certain cancer cells which allow the malignant cells to multiply and spread due to a change in the genetic make up of the cancer cell.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the proportion of participants with metastatic mucosal or acral/lentiginous melanoma who are alive and without disease progression at two months after beginning treatment with sunitinib.
* To determine the best overall response rate.

Secondary

* To determine the time to progression and overall survival.
* To correlate c-kit mutational status with response to therapy.
* To evaluate the use of FDG-PET scanning in determining early biologic response to therapy.
* To assess amplification of c-kit status through quantitative PCR and/or FISH and other related molecular pathway targets.

ELIGIBILITY:
Inclusion Criteria:

* History of primary mucosal or acral/lentiginous melanoma
* Histologically documented stage III unresectable or IV metastatic melanoma
* ECOG Performance Status 0,1 or 2
* Estimated life expectancy of 6 months or greater
* 18 years of age or older
* Lab values as outlined in protocol
* Tumor blocks or slides must be available of either primary or metastatic tumor site for c-kit mutation testing
* Negative pregnancy test within 48 hours of starting treatment
* At least one measurable site of disease as defined by at least 1cm in greatest dimension

Exclusion Criteria:

* Severe and/or uncontrolled medical disease
* Pregnant or nursing mothers
* Known brain metastasis. History of or known spinal cord compression, or carcinomatous meningitis, or evidence of symptomatic brain or leptomeningeal disease on screening CT or MRI scan
* Less than 5 years free of another primary malignancy except: if the other primary malignancy is not currently clinically significant nor requiring active intervention, or if other primary malignancy is a basal cell skin cancer or cervical carcinoma in situ
* Grade III/IV cardiac problems as defined by the New York Heart Association Criteria
* Ongoing cardiac dysrhythmias of grade 2 or greater, atrial fibrillation, QTc interval >450msec for males of >470 msec for females
* Hypertension that cannot be controlled by medication
* Any of the following within 12 months prior to starting treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism
* NCI CTCAE version 3.0 grade 3 hemorrhage within 4 weeks of starting the study treatment
* Concurrent treatment with warfarin
* Prior treatment with SU011248 or any other antiangiogenic agent
* No H2 blockers or proton pump inhibitors
* Known chronic liver disease
* Known HIV infection
* Previous radiotherapy to 25% or more of the bone marrow and/or radiation therapy within 4 weeks prior to study entry
* Major surgery within 4 weeks prior to study entry
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: F. Stephen Hodi, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Buchbinder EI, Sosman JA, Lawrence DP, McDermott DF, Ramaiya NH, Van den Abbeele AD, Linette GP, Giobbie-Hurder A, Hodi FS. Phase 2 study of sunitinib in patients with metastatic mucosal or acral melanoma. Cancer. 2015 Nov 15;121(22):4007-15. doi: 10.1002/cncr.29622. Epub 2015 Aug 11. PMID 26264378

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study, conducted at 7 medical centers, was activated on August 8, 2007 and closed on August 1, 2014. Patient enrollment to Cohort A occurred from September 2007 to January 2009 and Cohort B from March 2009 to June 2013.
Pre-assignment Details: The trial was amended in 2009 to revise sunitinib dosing due to difficulty with tolerability and evidence of progressive disease following treatment breaks. As such, there are two study cohorts: the first employing intermittent dosing of Sunitinib (Cohort A) and the second with continuous dosing (Cohort B).
Groups:
- Cohort A-Sunitinib Intermittent Dosing: Cohort A participants received 50 mg sunitinib orally daily for 4 weeks followed by a two-week break from treatment. These 6-week cycles would be repeated until progression or unacceptable toxicity up to 1 year.
- Cohort B-Sunitinib Continuous Dosing: Cohort B participants received 37.5 mg sunitinib daily on a continuous basis until progression or unacceptable toxicity up to 1 year.
Period: Overall Study
Arm/Group | Cohort A-Sunitinib Intermittent Dosing | Cohort B-Sunitinib Continuous Dosing
Started | 21 | 31
Completed | 0 (Since treatment duration was not fixed, patients were not considered to have completed treatment.) | 0 (Since treatment duration was not fixed, patients were not considered to have completed treatment.)
Not Completed | 21 | 31
Not completed — Adverse Event | 0 | 6
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Progressive Disease | 17 | 19
Not completed — Intercurrent Illness | 1 | 2
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of treated patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A-Sunitinib Intermittent Dosing | Cohort B-Sunitinib Continuous Dosing | Total
Number analyzed (Participants) | 21 | 31 | 52
Age, Continuous [Median (Full Range); unit: years] | 63 [38 to 80] | 63 [40 to 86] | 63 [38 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 20 | 30
  Male | 11 | 11 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 21 | 28 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 31 | 52

OUTCOME MEASURES:

1. Primary Outcome: 2-month Progression-free Survival Rate
Description: 2-month progression-free survival rate was defined as the proportion of patients absent death or progression based on Response Evaluation Criteria In Solid Tumors Criteria (RECIST) before 2 months. Per RECIST 1.0 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease was evaluated radiologically at baseline and every 8 weeks on treatment; Treatment continued for 12 months unless disease progression or unacceptable toxicity. Relevant for this endpoint was disease status at 2 months.
Population: The analysis dataset is comprised of treated patients.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Cohort A-Sunitinib Intermittent Dosing | Cohort B-Sunitinib Continuous Dosing
Number analyzed (Participants) | 21 | 31
proportion of patients | .52 [.30 to .74] | .52 [.33 to .70]

2. Secondary Outcome: Best Overall Response Rate
Description: The best overall response rate was defined as achieving partial response (PR) or complete response (CR) on treatment based on RECIST 1.0 criteria. Per RECIST 1.0 for target lesions, CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. To be assigned a status of CR or PR, changes in tumor measurements must be confirmed by repeat assessments performed no fewer than 4 weeks after the response criteria are first met. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Disease was evaluated radiologically at baseline and every 8 weeks on treatment. Mean treatment duration was 3 cycles (Cohort A/B mean 2/3 cycles). The range of treatment duration overall was 1-11 cycles.
Population: The analysis dataset is comprised of treated patients.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort A-Sunitinib Intermittent Dosing | Cohort B-Sunitinib Continuous Dosing
Number analyzed (Participants) | 21 | 31
proportion of participants | 0.095 [0.012 to 0.304] | 0.065 [0.0078 to 0.214]

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from study entry to death or date last known alive.
Time Frame: Patients were followed long-term every 3 months until first progression, death or lost to follow-up. Median survival follow-up was 6.7 months (range 0.8-47.3 months; Cohort A/B median 7.7 m/ 6.2 m).
Population: The analysis dataset is comprised of treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A-Sunitinib Intermittent Dosing | Cohort B-Sunitinib Continuous Dosing
Number analyzed (Participants) | 21 | 31
months | 7.7 [6.9 to 14.9] | 6.8 [5.2 to 9.6]

4. Secondary Outcome: Time to Progression
Description: Time to progression based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) requiring removal from the study. Per RECIST 1.0 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease was evaluated radiologically at baseline and every 8 weeks on treatment and long-term every 3 months until first progression, death or lost to follow-up. Mean treatment duration was 3 cycles (range 1-11; Cohort A/B mean 2/3 cycles).
Population: The analysis dataset is comprised of treated patients. The majority of patients were off-treatment due to disease progression and thus the relevant observation time frame for this outcome is time on treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A-Sunitinib Intermittent Dosing | Cohort B-Sunitinib Continuous Dosing
Number analyzed (Participants) | 21 | 31
months | 2.7 [1.7 to 4.1] | 3.6 [1.7 to 3.9]

ADVERSE EVENTS:
Time Frame: AE assessment was ongoing from the start of study drug and up to day 30 post-treatment.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv3. Other AEs were defined as events with treatment-attribution of possible, probable or definite and grades 1 or 2 per CTCAEv3.
Arm/Group | Cohort A-Sunitinib Intermittent Dosing | Cohort B-Sunitinib Continuous Dosing
Serious Adverse Events (participants affected / at risk) | 10/21 | 13/31
Other Adverse Events (participants affected / at risk) | 19/21 | 24/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A-Sunitinib Intermittent Dosing (N=21) | Cohort B-Sunitinib Continuous Dosing (N=31)
ALT, SGPT (Investigations) | 1 | 0
Amylase (Investigations) | 2 | 2
AST, SGOT (Investigations) | 1 | 0
Death - sudden death (General disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 0 | 2
Hemoglobin (Blood and lymphatic system disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 1
Infection w/ gr3-4 neut, nose (Infections and infestations) | 0 | 1
Leukocytes (Investigations) | 1 | 3
Lipase (Investigations) | 2 | 3
Lymphopenia (Investigations) | 1 | 3
Neutrophils (Investigations) | 0 | 3
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Platelets (Investigations) | 0 | 3
Stomach, hemorrhage (Gastrointestinal disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A-Sunitinib Intermittent Dosing (N=21) | Cohort B-Sunitinib Continuous Dosing (N=31)
Abdomen, pain (Gastrointestinal disorders) | 1 | 0
Alkaline phosphatase (Investigations) | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
ALT, SGPT (Investigations) | 2 | 3
Amylase (Investigations) | 3 | 3
Anorexia (Metabolism and nutrition disorders) | 6 | 5
Ascites (non-malignant) (Gastrointestinal disorders) | 0 | 1
AST, SGOT (Investigations) | 4 | 7
Bicarbonate (Metabolism and nutrition disorders) | 1 | 0
Bronchopulmonary, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cardiac/heart, pain (Cardiac disorders) | 1 | 0
Cardiac (Cardiac disorders) | 1 | 0
CD4 (Investigations) | 0 | 1
Confusion (Psychiatric disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 5 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Creatinine (Investigations) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 4 | 11
Distention/bloating, abdominal (Gastrointestinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 5
Dysphagia (Gastrointestinal disorders) | 2 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Edema head and neck (General disorders) | 1 | 0
Edema limb (General disorders) | 2 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Fatigue (General disorders) | 14 | 12
Fever w/o neutropenia (General disorders) | 2 | 1
GI-other (Gastrointestinal disorders) | 5 | 1
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 0 | 6
Head/headache (Nervous system disorders) | 2 | 0
Hematologic (Blood and lymphatic system disorders) | 1 | 1
Hemoglobin (Blood and lymphatic system disorders) | 4 | 7
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Hepatic (Hepatobiliary disorders) | 1 | 0
Hyopthyroidism (Endocrine disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 3 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 1
Hyponatremia (Metabolism and nutrition disorders) | 3 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 3
Hypotension (Vascular disorders) | 1 | 0
Incontinence, anal (Gastrointestinal disorders) | 1 | 0
Infection Gr0-2 neut, skin (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Joint, pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Leukocytes (Investigations) | 10 | 11
Lipase (Investigations) | 4 | 2
Lymphopenia (Investigations) | 3 | 2
Muco/stomatitis (symptom) esophagus (Gastrointestinal disorders) | 0 | 1
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 3 | 3
Muco/stomatitis (symptom) stomach (Gastrointestinal disorders) | 0 | 1
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 1 | 2
Nail changes (Skin and subcutaneous tissue disorders) | 2 | 0
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 8 | 7
Neurologic-other (Nervous system disorders) | 2 | 1
Neuropathy-sensory (Nervous system disorders) | 0 | 1
Neutrophils (Investigations) | 10 | 6
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Ocular-other (Eye disorders) | 1 | 0
Odor (patient odor) (Skin and subcutaneous tissue disorders) | 1 | 0
Optic disc edema (Eye disorders) | 1 | 0
Oral cavity, pain (Gastrointestinal disorders) | 2 | 2
Pain-other (General disorders) | 3 | 1
Platelets (Investigations) | 9 | 10
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 | 2
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 | 1
Renal/GU (Renal and urinary disorders) | 0 | 1
Retinopathy (Eye disorders) | 0 | 1
Rigors/chills (General disorders) | 1 | 0
Skin (Skin and subcutaneous tissue disorders) | 3 | 1
Stomach, pain (Gastrointestinal disorders) | 2 | 0
Sweating (Skin and subcutaneous tissue disorders) | 2 | 0
Taste disturbance (Nervous system disorders) | 9 | 8
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Urinary frequency/urgency (Renal and urinary disorders) | 1 | 1
Vagina, pain (Reproductive system and breast disorders) | 1 | 0
Vaginal mucositis (Reproductive system and breast disorders) | 1 | 0
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Vomiting (Gastrointestinal disorders) | 5 | 5
Weight loss (Investigations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No